CLINICAL TRIAL: NCT03250741
Title: Effects of Dopaminergic Therapy in Patients With Alzheimer's Disease: a Phase II 24-week, Randomized, Double-blind Placebo Controlled Study.
Brief Title: Effects of Dopaminergic Therapy in Patients With Alzheimer's Disease
Acronym: DOPAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giacomo Koch, PI, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2015-002965-43
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer Disease
Keywords: Rotigotine; Dopamine
MeSH Terms: conditions — Alzheimer Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (2):
- Rotigotine 4 mg (Active Comparator): Rotigotine transdermal patches 4 mg
  Interventions: Drug: Rotigotine transdermal patch
- Placebo (Placebo Comparator): Placebo transdermal patches
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rotigotine transdermal patch — Rotigotine transdermal patches 4mg/24hr
  Other Names: ROTIGOTINE
  Arms: Rotigotine 4 mg
Other: Placebo — Placebo transdermal patches of the same size as for Rotigotine transdermal patches
  Other Names: Placebo transdermal patch
  Arms: Placebo

SUMMARY:
This is phase IIa 24-week, prospective, randomized, double-blind placebo controlled study. The study is designed to evaluate the efficacy, safety, and tolerability of transdermal patch of Rotigotine (RTG) versus placebo (PLC) as add-on therapy with AChEI in patients with mild AD according to the consensus diagnostic criteria and MMSE score of ≥18 and ≤24 at screening. Two groups of patients with mild AD will be involved (50 patients each). One group will be assigned to treatment with RTG 4 mg and the other one to PLC as add on to AChEI therapy (Rivastigmine). Clinical and neurophysiological measurements will be collected before and after drug administration.

DETAILED DESCRIPTION:
The current study has the ambition to provide first time evidence that dopaminergic stimulation may have a clinical impact in patients with mild AD.

Cognitive Assessment: Before and after the 24 weeks of treatment the ADAS-Cog, ADCS-ADL and the Frontal assessment battery (FAB) will be administered. FAB will be performed to measure changes in frontal executive functions (Apollonio et al, 2005) .

Neurophysiological investigations will be performed to identify quantifiable biomarkers underlying the effects induced by dopamine agonist on the neurodegenerative brain. The application of recent neurophysiological tools, such as the combined use of transcranial magnetic stimulation (TMS) during electroencephalography (EEG) will allow to measure how dopamine agonists are able to modulate the cortical activity of the prefrontal cortex in AD patients (Kähkönen et al., 2005; Julkunen et al., 2008), likely trough DA terminals originating from the ventral tegmental nucleus, defining the neurophysiological biomarkers of clinical improvement For EEG-TMS recordings, a TMS-compatible EEG equipment will be used for recording EEG activity from the scalp (BrainAmp 32MRplus, BrainProducts). The EEG will be continuously acquired from 64 scalp sites positioned according to the 10-20 International System. To precisely position the coil over the cortical sites across different sessions, a neuronavigation system (Softaxic, E.M.S.) will be used. Neurophysiological changes induced by dopamine-agonist will be indexed by the following measures: corticospinal excitability, cortical reactivity, connectivity and plasticity. Specifically, the cortical reactivity and cortico-cortical connectivity will be evaluated respectively over the prefrontal cortex and between connected areas. We will employ TMS-evoked cortical responses (i.e., TEPs) as a novel probe of dopamine-agonist induced cortical excitability changes (Ilmoniemi et al., 1997; Komssi and Kahkonen, 2006; Julkunen et al., 2008; Miniussi and Thut, 2009; Miniussi et al., 2012; Premoli et al., 2014). To reach this aim, TEPs will serve as markers of left prefrontal cortex (PFC) reactivity whereas the spreading of their cortical activation will serve as an index of connectivity between targeted cortex and functionally connected areas underlying frontal cognitive network.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (or if applicable the legally acceptable representative if different from the responsible caregiver) and the responsible caregiver have signed the Informed Consent Form.
2. The patient has probable AD, diagnosed according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
3. The patient is a man or woman, aged ≤ 85 years.
4. The patient has a Clinical Dementia Rating (CDR) total score of 0.5 or 1 (mild) and MMSE score of 20-26 (inclusive) at Screening.
5. Has at least one identified adult caregiver who is able to provide meaningful assessment of changes in subject behavior and function over time and provide information on safety and tolerability, and is able to verify daily compliance with study drug
6. The patient has been treated with acetylcholinesterase inhibitor (AChEI), i.e., donepezil, galantamine, or rivastigmine, at the time of Screening

   * For at least 3 months
   * The current dosage regimen and must have remained stable for ≥ 8 weeks
   * It must be planned that the dosage regimen will remain stable throughout participation in the study

Exclusion Criteria:

1. Significant neurodegenerative disorder of the central nervous system other than Alzheimer's disease, e.g., Lewy body dementia, Parkinson's disease, multiple sclerosis, progressive supranuclear palsy, hydrocephalus, Huntington's disease, any condition directly or indirectly caused by Transmissible Spongiform Encephalopathy (TSE), Creutzfeldt-Jakob Disease (CJD), variant Creutzfeldt-Jakob Disease (vCJD), or new variant Creutzfeldt-Jakob Disease (nvCJD)
2. The patients has history of seizure (with the exception of febrile seizures in childhood)
3. Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM IV-TR) criteria met for any of the following within specified period:

   * Major depressive disorder (current)
   * Schizophrenia (lifetime)
   * Other psychotic disorders, bipolar disorder, or substance (including alcohol) related disorders (within the past 5 years)
4. Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MR imaging.
5. Evidence of clinically significant disease including but not limited to pulmonary, gastrointestinal, renal, hepatic, endocrine, cardiovascular or metabolic disorder (Patients with controlled diabetes, or hypertension, or complete/partial right bundle branch block may be included in the study).
6. Treatment currently or within 6 months before Baseline with any of the following medications:

   * Typical and atypical antipsychotics (i.e. Clozapine, Olanzapine)
   * Antiparkinson agents (e.g., levodopa, dopamine agonists, COMT inhibitors, amantadine, monoamine oxidase B inhibitors, anticholinergics etc)
   * Carbamazepine, Primidone, Pregabalin, Gabapentin
   * Memantine

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Global cognition | change from baseline to Week 24
  Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)

SECONDARY OUTCOMES:
Frontal cognitive functions | change from baseline to Week 24
  Frontal assessment battery (FAB)
Activities of daily living | change from baseline to Week 24
  Alzheimer's disease Cooperative Study - Activities of Daily Living (ADCS-ADL)
Neurophysiological markers of cortical activity | change from baseline to Week 24
  TEP amplitude over the PFC
Neuropsychiatric evaluation | change from baseline to Week 24
  Neuropsychiatric Inventory (NPI)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Martorana, MD, PhD, Study Director — University of Rome Tor Vergata; Giacomo Koch, MD, PhD, Principal Investigator — Santa Lucia Foundation IRCCS
Locations (1):
- Santa Lucia Foundation, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martorana A, Di Lorenzo F, Esposito Z, Lo Giudice T, Bernardi G, Caltagirone C, Koch G. Dopamine D(2)-agonist rotigotine effects on cortical excitability and central cholinergic transmission in Alzheimer's disease patients. Neuropharmacology. 2013 Jan;64:108-13. doi: 10.1016/j.neuropharm.2012.07.015. Epub 2012 Aug 1. PMID 22863599
- [Result] Martorana A, Koch G. "Is dopamine involved in Alzheimer's disease?". Front Aging Neurosci. 2014 Sep 25;6:252. doi: 10.3389/fnagi.2014.00252. eCollection 2014. PMID 25309431
- [Result] Koch G, Di Lorenzo F, Bonni S, Giacobbe V, Bozzali M, Caltagirone C, Martorana A. Dopaminergic modulation of cortical plasticity in Alzheimer's disease patients. Neuropsychopharmacology. 2014 Oct;39(11):2654-61. doi: 10.1038/npp.2014.119. Epub 2014 May 26. PMID 24859851
- [Derived] Koch G, Motta C, Bonni S, Pellicciari MC, Picazio S, Casula EP, Maiella M, Di Lorenzo F, Ponzo V, Ferrari C, Scaricamazza E, Caltagirone C, Martorana A. Effect of Rotigotine vs Placebo on Cognitive Functions Among Patients With Mild to Moderate Alzheimer Disease: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jul 1;3(7):e2010372. doi: 10.1001/jamanetworkopen.2020.10372. PMID 32667654